CLINICAL TRIAL: NCT04712227
Title: Can the Ratio of Chin-neck Circumference and Neck Circumference to Chin-neck Circumference Predict Difficult Intubation in Obese Patients?
Acronym: intubation
Status: Completed | Type: Observational
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, adem selvi, uzman doktor, Kecioren Education and Training Hospital
Other Study IDs: adem obez havayolu
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Difficult Airway Intubation; Obesity Adult Onset
Keywords: neck circumference / chin-nape circumference; chin-nape circumference; difficult airway; obesity
MeSH Terms: conditions — Obesity | interventions — Intubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- difficult intubation: patients with a difficult intubation score of 5 or more
  Interventions: Other: intubation
- easy intubation: patients with difficult intubation score less than 5
  Interventions: Other: intubation
- difficult mask ventilation: group 3 and 4 by han mask ventilation grouping
  Interventions: Other: mask ventilation
- easy mask ventilation: group 1 and 2 according to han mask ventilation grouping
  Interventions: Other: mask ventilation

INTERVENTIONS:
Other: intubation — intubation
  Groups: difficult intubation; easy intubation
Other: mask ventilation — mask ventilation
  Groups: difficult mask ventilation; easy mask ventilation

SUMMARY:
Importance and Purpose of the Study: Proper management of the difficult airway is an important part of preventing anesthesia-related mortality and morbidity. Difficult airways, characterized by both difficult mask ventilation and difficult intubation, are common in obese patients. Many studies have shown an association between obesity or morbid obesity and difficult intubation. We thought that in obese patients, increased subcutaneous fat tissue in the nape of the neck may restrict the head extension and cause difficult intubation and difficult mask ventilation, and the increase in the chin-nape circumference may predict difficult intubation and difficult mask ventilation. We also predicted that the ratio of neck circumference to chin-nape circumference might predict difficult intubation and difficult mask ventilation.

Materials and Methods: After the approval of the ethics committee, obese patients who require tracheal intubation, undergo elective surgery, over the age of 18, with a body mass index (BMI) of more than 30 were evaluated. Patients with cervical spine anomaly, emergency procedures, known history of difficult intubation or upper respiratory tract disease, and planned awake intubation were excluded from the study. Mallampati score, mouth opening, upper lip bite test, distance between incisors, thyromental distance, sternomental distance and thyromental height were recorded. Using a tape measure, the neck circumference from the thyroid cartilage level and the chin-neck circumference from the mentum level were measured with the patient in a neutral position. The ratio of neck circumference to thyromental distance and the ratio of neck circumference to chin-nape circumference were calculated from these measurements. Mask ventilation was graded according to the method described by Han et al. After adequate muscle relaxation was achieved, tracheal intubation was performed with an appropriately sized Macintosh blade using direct laryngoscopy. Difficult intubation evaluation was performed using the Difficult Intubation Scale (IDS) based on seven variables.

Results: A statistically significant relationship was found between difficult intubation and the distance between incisors, neck circumference, neck circumference / thyromental distance, neck circumference / sternomental distance, and chin-nape circumference. In the multivariate regression analysis performed with these parameters, the distance between the incisors was <4.85 cm and the neck circumference> 41.5 cm was found to be independent risk factors for difficult intubation. A statistically significant relationship was found between difficult mask ventilation and age, male gender, OSAS, neck circumference, neck circumference / thyromental distance, neck circumference / sternomental distance, neck circumference / chin-nape circumference and chin-nape circumference. In the multivariate regression analysis performed with these parameters, it was determined that male gender and neck circumference thicker than 45.5 cm were independent risk factors for difficult mask ventilation.

Conclusion: The ratio of neck circumference to chin-nape circumference and chin-nape circumference are successful in predicting difficult mask ventilation in obese patients. While chin-nape circumference is successful in predicting difficult intubation in obese patients, neck circumference / chin-nape circumference is unsuccessful.

ELIGIBILITY:
Inclusion Criteria: Patients who will be operated under general anesthesia with endotracheal intubation, aged 18 years and over, with body mass index (BMI≥30) and ASA 1-3

Exclusion Criteria:Patients with cervical spine anomalies, emergency procedures, known difficult intubation history and awake intubation plan, and those with beard were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will be operated under general anesthesia with endotracheal intubation, aged 18 years and over, with body mass index (BMI≥30) and ASA 1-3
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Parameters associated with difficult intubation in obese patients | always
  mallampati score, cormack-lehane score, distance between incisors, neck circumference, ratio of neck circumference to thyromental distance, ratio of neck circumference to sternomental distance and chin-nape circumference

SECONDARY OUTCOMES:
parameters associated with difficult mask ventilation in obese patients | always
  age, gender, OSAS, neck circumference, chin-nape circumference, ratio of neck circumference to chin-nape circumference, ratio of neck circumference to thyromental distance, and ratio of neck circumference to sternomenal distance

CONTACTS AND LOCATIONS:
Overall Officials: adem selvi, uzman dr., Principal Investigator — sorumlu araştırmacı
Locations (1):
- Keçiören training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
everything
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months
Access Criteria: difficult airway obesity

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04712227/Prot_SAP_000.pdf